CLINICAL TRIAL: NCT05302713
Title: Evaluating Changes in Quality of Life and Epigenetic Methylation From Antiorbital Ionic Calcium in Older Adults With Chronic Conditions
Brief Title: Antiorbital Calcium in Chronic Conditions
Acronym: AntiAFib
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Ryan Bradley, Director of Research, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RB121521
Record Dates: First submitted 2022-03-16; First posted 2022-03-31 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; calcium; supplements; antiorbital ionic calcium; quality of life
MeSH Terms: conditions — Atrial Fibrillation | interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to take either an ionic calcium (IC) supplement or calcium carbonate (CC) supplement for 12 weeks. At the 12 week time point, all participants, whether having taken IC or CC for the first 12 weeks, will take the IC supplement for the final 12 weeks of the study in an open label fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ionic Calcium (Experimental): Ionic calcium (IC) is a calcium in a free ionic state. Participants will be instructed to take 8mg of IC/60kg body weight dissolved into approximately 500ml of purified water. Participants will titrate their dose at the start of the study as follows: days 1-3: 1 dose per day 30 min prior to a meal; Days 4-6: twice per day, 30 minutes before meals; from day seven onward, the full dosage of three times per day, 30 minutes before meals.
  Interventions: Dietary Supplement: Ionic Calcium
- Calcium Carbonate (Active Comparator): Participants will be instructed to take 8mg of calcium carbonate/60kg body weight dissolved into approximately 500ml of purified water. Participants will titrate their dose at the start of the study as follows: days 1-3: 1 dose per day 30 min prior to a meal; Days 4-6: twice per day, 30 minutes before meals; from day seven onward, the full dosage of three times per day, 30 minutes before meals.
  Interventions: Dietary Supplement: Calcium Carbonate

INTERVENTIONS:
Dietary Supplement: Ionic Calcium — Ionic calcium (IC), a calcium in a free ionic state (i.e., non-protein bound), is purported to improve calcium uptake and homeostasis leading to improved cellular signaling that may have been disrupted through environmental and lifestyle stressors.
  Arms: Ionic Calcium
Dietary Supplement: Calcium Carbonate — Calcium carbonate supplementation in a solution identical in appearance, consistency, and taste to the intervention supplement.
  Arms: Calcium Carbonate

SUMMARY:
The purpose of this study is to determine the mechanistic effects of an ionic calcium supplement in adults with atrial fibrillation, osteoarthritis, and hypertension. The study aims to determine if ionic calcium supplementation affects quality of life, rate of biological aging, bone densitometry, and blood biomarkers of bone metabolism over a six month period compared to non-ionic calcium comparator supplement.

ELIGIBILITY:
Inclusion criteria:

* Adults 55-75 years of age
* Active diagnosis of one of the following conditions:
* Stage 1 Hypertension with Non-valvular Atrial Fibrillation (AF) - including paroxysmal, persistent, or long-standing persistent AF with typical electrocardiographic characteristics (i.e., absence of identifiable p-waves with irregularly irregular ventricular rate) without known complications, heart disease, or congenital heart defects (e.g., rapid ventricular rate, recent myocardial infarction, heart failure, stroke, cardiomyopathy, etc.), self-reported but previously diagnosed by a healthcare professional;
* Stage 1 Hypertension (systolic blood pressure of 130-139, diastolic blood pressure of 80-89), self-reported but previously diagnosed by a healthcare professional;
* or, Osteoarthritis, self-reported but previously diagnosed by a healthcare professional.
* If diagnosed with AF, a European Heart Rhythm Association (EHRA) score of 2b or greater (i.e. Normal daily activity not affected by symptoms related to AF, but patient troubled by symptoms).
* On a stable dose of all medications prior to study entry (i.e., consistent dose for a minimum of three months)
* Willing to be randomized to take daily ionized calcium as a dietary supplement or placebo over the 24-week study period
* On a stable dose of dietary supplements for at least one month prior to enrollment
* Willing to avoid initiation of new supplements and/or medications unless otherwise indicated by a healthcare professional
* Willing to have blood drawn on 6 occasions, and fast for 10-12 hours before blood draws, over the study period
* Willing to have desktop ultrasound of wrist done on 3 occasions.
* Able to communicate via email, complete computer-administered questionnaires, and to read and write in English.
* Must be able to provide written informed consent
* Non-smokers (including tobacco and cannabis products, combusted or vaporized)
* Approved to be eligible for study participation at the discretion of the Principal Investigators, after review of the Formal Eligibility Screen results.
* Willing to avoid taking dietary supplements containing the following ingredients for the 24 weeks of study involvement: additional supplemental calcium in any form, vitamin D, vitamin K, selenium, magnesium, or zinc.

Exclusion criteria:

* Individuals with a current or past diagnosis of permanent AF
* Individuals with any thyroid or parathyroid disorders, or current use of thyroid medication for any reason.
* Individuals with chronic kidney or liver disease, cancer, colorectal disease, and "other rare disorders".
* Individuals with a current diagnosis of Congestive Heart Failure (CHF).
* Individuals with a current or past diagnosis of Traumatic Brain Injury (TBI), thromboembolism, or Cerebrovascular Accident (CVA)/Stroke.
* Use of dihydropyridine or non-dihydropyridine calcium channel blockers for any reason
* If diagnosed with atrial fibrillation, not on a stable dose of anti-coagulant or anti-platelet prescription medications (i.e., consistent dose for a minimum of three months)
* Abnormalities in coagulation studies (e.g., INR ≤ 2 or ≥ 3.0) or hypercalcemia at the clinical screening visit.
* Blood pressure ≥ 140/90 mmHg at the clinical screening visit.
* Current involvement or within 14 days prior to screening of a significant diet or weight loss program (such as NutriSystem, Jenny Craig, Atkin's or other low-carb diet programs) or very low-calorie liquid diet programs (such as Optifast, Medifast, and/or HMR)
* Hospitalization (for any reason other than a scheduled medical procedure unrelated to atrial fibrillation, hypertension, or osteoarthritis) within 3 months prior to screening
* Cardiac surgery within 3 months prior to screening
* Malignancy within the last 5 years (with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix)
* Are allergic to corn.
* Women who are lactating, pregnant or planning pregnancy within the next six months
* Intake of ≥ 2 standardized alcohol-containing beverages per day, 14 per week, or ≥4 in any single day within the past 14 days.
* Women who experience menstrual periods, who are sexually active and are unwilling to use an appropriate form of contraception during the duration of the trial.
* Smoking tobacco or nicotine products (combusted or vaporized)
* Use of illicit drugs/substances (such as but not limited to cocaine, phencyclidine (PCP), and methamphetamine) within 14 days of screening
* Currently participating in another interventional research study, or participated in another interventional research study within 14 days of screening
* Do not have an active primary care provider or specialist (i.e., cardiologist, rheumatologist, orthopedist, etc.) managing their atrial fibrillation, hypertension, or osteoarthritis.
* Current use of: dietary supplements or medications utilized for chelation purposes (i.e., ethylenediaminetetraacetic acid; EDTA), or of chemotherapeutic agents.
* MoCA score of 16 or less upon screening.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Biological Aging | Baseline
  Dunedin Pace of Aging Calculated objective measure of the rate of epigenetic aging
Rate of Biological Aging | Week 12
  Dunedin Pace of Aging Calculated objective measure of the rate of epigenetic aging
Rate of Biological Aging | Week 24
  Dunedin Pace of Aging Calculated objective measure of the rate of epigenetic aging
Patient Reported Outcomes Measurement Information system-29 Physical Function Sub-domain | Baseline
  Quality of Life
Patient Reported Outcomes Measurement Information system-29 Physical Function Sub-domain | Week 2
  Quality of Life
Patient Reported Outcomes Measurement Information system-29 Physical Function Sub-domain | Week 6
  Quality of Life
Patient Reported Outcomes Measurement Information system-29 Physical Function Sub-domain | Week 12
  Quality of Life
Patient Reported Outcomes Measurement Information system-29 Physical Function Sub-domain | Week 24
  Quality of Life

SECONDARY OUTCOMES:
Changes in Systolic and Diastolic Blood Pressure | Baseline
  Objective measure of blood pressure
Changes in Systolic and Diastolic Blood Pressure | Week 2
  Objective measure of blood pressure
Changes in Systolic and Diastolic Blood Pressure | Week 6
  Objective measure of blood pressure
Changes in Systolic and Diastolic Blood Pressure | Week 12
  Objective measure of blood pressure
Changes in Systolic and Diastolic Blood Pressure | Week 24
  Objective measure of blood pressure
Changes in Cognition | Baseline
  MoCA Assessment Score
Changes in Cognition | Week 6
  MoCA Assessment Score
Changes in Cognition | Week 12
  MoCA Assessment Score
Changes in Cognition | Week 24
  MoCA Assessment Score
Changes in Mood | Baseline
  Patient Health Questionnaire-9 Score
Changes in Mood | Week 2
  Patient Health Questionnaire-9 Score
Changes in Mood | Week 6
  Patient Health Questionnaire-9 Score
Changes in Mood | Week 12
  Patient Health Questionnaire-9 Score
Changes in Mood | Week 24
  Patient Health Questionnaire-9 Score
Changes in Anxiety | Baseline
  Generalized Anxiety Disorder-7 Score
Changes in Anxiety | Week 2
  Generalized Anxiety Disorder-7 Score
Changes in Anxiety | Week 6
  Generalized Anxiety Disorder-7 Score
Changes in Anxiety | Week 12
  Generalized Anxiety Disorder-7 Score
Changes in Anxiety | Week 24
  Generalized Anxiety Disorder-7 Score
Changes in Pain and Disability | Baseline
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score
Changes in Pain and Disability | Week 2
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score
Changes in Pain and Disability | Week 6
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score
Changes in Pain and Disability | Week 12
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score
Changes in Pain and Disability | Week 24
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score

OTHER OUTCOMES:
Coronary Artery Calcium Score | Week 12
  Composite Coronary Artery Calcium Score
Coronary Artery Calcium Score | Week 24
  Composite Coronary Artery Calcium Score
Ultrasonometer Bone Densitometry | Week 12
  Bone density T score resulting from ultrasound
Ultrasonometer Bone Densitometry | Week 24
  Bone density T score resulting from ultrasound
Activated Partial Thromboplastin Time | Week 2
  Measure of blood coagulation
Activated Partial Thromboplastin Time | Week 6
  Measure of blood coagulation
Activated Partial Thromboplastin Time | Week 12
  Measure of blood coagulation
Activated Partial Thromboplastin Time | Week 24
  Measure of blood coagulation
Prothrombin Time | Week 2
  Measure of blood coagulation
Prothrombin Time | Week 6
  Measure of blood coagulation
Prothrombin Time | Week 12
  Measure of blood coagulation
Prothrombin Time | Week 24
  Measure of blood coagulation
Internationalized Normalized Ratio | Week 2
  Measure of blood coagulation
Internationalized Normalized Ratio | Week 6
  Measure of blood coagulation
Internationalized Normalized Ratio | Week 12
  Measure of blood coagulation
Internationalized Normalized Ratio | Week 24
  Measure of blood coagulation
Thrombin Time | Week 12
  Measure of blood coagulation
Thrombin Time | Week 24
  Measure of blood coagulation
Concentration of Serum Calcium (ionic) | Week 12
  Measure of non-protein bound calcium concentration in the serum
Concentration of BUN (serum) | Week 2
  Measure of renal function and protein turnover
Concentration of BUN (serum) | Week 6
  Measure of renal function and protein turnover
Concentration of BUN (serum) | Week 12
  Measure of renal function and protein turnover
Concentration of BUN (serum) | Week 24
  Measure of renal function and protein turnover
Concentration of Creatinine (serum) | Week 2
  Measure of renal function
Concentration of Creatinine (serum) | Week 6
  Measure of renal function
Concentration of Creatinine (serum) | Week 12
  Measure of renal function
Concentration of Creatinine (serum) | Week 24
  Measure of renal function
Glomerular Filtration Rate, estimated (eGFR) | Week 2
  Measure of renal function
Glomerular Filtration Rate, estimated (eGFR) | Week 6
  Measure of renal function
Glomerular Filtration Rate, estimated (eGFR) | Week 12
  Measure of renal function
Glomerular Filtration Rate, estimated (eGFR) | Week 24
  Measure of renal function
Concentration of Alanine aminotransferase (serum) | Week 2
  Measure of liver function
Concentration of Alanine aminotransferase (serum) | Week 6
  Measure of liver function
Concentration of Alanine aminotransferase (serum) | Week 12
  Measure of liver function
Concentration of Alanine aminotransferase (serum) | Week 24
  Measure of liver function
Concentration of Aspartate aminotransferase (serum) | Week 2
  Measure of liver function
Concentration of Aspartate aminotransferase (serum) | Week 6
  Measure of liver function
Concentration of Aspartate aminotransferase (serum) | Week 12
  Measure of liver function
Concentration of Aspartate aminotransferase (serum) | Week 24
  Measure of liver function
Concentration of Thyroid Stimulating Hormone | Week 2
  Measure of thyroid activity
Concentration of Thyroid Stimulating Hormone | Week 6
  Measure of thyroid activity
Concentration of Thyroid Stimulating Hormone | Week 12
  Measure of thyroid activity
Concentration of Thyroid Stimulating Hormone | Week 24
  Measure of thyroid activity
Concentration of Calcitonin | Week 12
  Measure of bone formation
Concentration of Osteocalcin | Week 12
  Measure of bone formation
Concentration of Bone-Specific Alkaline Phosphatase | Week 12
  Measure of bone turnover
Concentration of Procollagen Type I Intact N Terminal Propeptide (PINP) | Week 12
  Measure of bone formation
Concentration of Collagen Type I C-Telopeptide (CTx) | Week 12
  Measure of bone resorption

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, Principal Investigator — National University of Natural Medicine
Locations (1):
- Helfgott Research Institute, Portland, Oregon, United States